CLINICAL TRIAL: NCT00512590
Title: Effects of Guided Imagery on Pain, Distress, Functional Status and Self-Efficacy in Hispanics Diagnosed With Fibromyalgia
Brief Title: Pilot Study: Relaxation and Guided Imagery in Hispanic Persons Diagnosed With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: Sigma Theta Tau International Honor Society of Nursing (Other); American Nurses Foundation (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Menzies-1
Record Dates: First submitted 2007-08-03; First posted 2007-08-07 (Estimated); Last update posted 2007-08-07 (Estimated); Status verified 2007-08

CONDITIONS: Fibromyalgia; Pain; Functional Status; Self-Efficacy; Distress
Keywords: fibromyalgia; relaxation; imagery; pain; functional status; self efficacy; minority health
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Imagery, Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental)
  Interventions: Behavioral: Relaxation and Guided Imagery

INTERVENTIONS:
Behavioral: Relaxation and Guided Imagery — The intervention consisted of 3 relaxation and guided imagery audiotapes used in a proscribed order for 6 weeks and used in any order for weeks 7 through 10.
  Protocol: Tape 1: Basic Relaxation used for weeks 1 and 2. Tape 2: Pleasant Scene Imagery to elicit sensory involvement for enhanced sense of overall well-being; used for weeks 3 and 4. Tape 3: End-State Imagery designed to facilitate improved symptom management; used for weeks 5 and 6. Any of the tapes used as often as desired but at least once daily for weeks 7 to 10.

SUMMARY:
The purpose of this pilot study was to test the effects of a 10-week relaxation and guided imagery intervention on pain perception, functional status, self-efficacy and levels of distress in Hispanic adults diagnosed with fibromyalgia.

DETAILED DESCRIPTION:
Fibromyalgia (FM), a chronic widespread pain condition with an unknown pathogenesis and no known cure, affects 2 to 4 million persons in the adult US population. One of the most common conditions seen in rheumatology clinics world wide, including the US, Mexico, and Spain, FM is accompanied by various co-occurring symptoms such as fatigue, disturbed sleep, stiffness and depression. While studies of fibromyalgia in Hispanics have been reported in Spain, Brazil and Argentina, very few such studies have been reported in the United States. This gap exists despite data indicating that there are a reported 16 million Hispanics with rheumatic diseases in the US and that Hispanics (self-identified) form the fastest growing minority group in this country.

ELIGIBILITY:
Inclusion Criteria:

* ages 18 and older
* diagnosis of fibromyalgia based on the American College of Rheumatology criteria and documented by the patient's primary physician
* a minimum of a 6th grade education level
* an ability to understand and sign the consent form and understand and complete the intervention (pencil and paper) assignments.

Exclusion Criteria:

* presence of other systemic rheumatologic conditions such as rheumatoid arthritis, lupus, and/or Sjogren's Disease
* adequate functional status as indicated by a Fibromyalgia Impact Questionnaire score < 20
* inadequate cognitive status as evidenced by a Mini-Mental State Exam score < 25
* history of epilepsy
* major communicative disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2005-04; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Pain as measured by Short-Form McGill Pain Questionnaire | 10 weeks

SECONDARY OUTCOMES:
Functional Status as measured by the Fibromyalgia Impact Questionnaire | 10 weeks
Self-Efficacy as measured by the Arthritis Self-Efficacy Scale adapted for FM | 10 weeks
Distress as measured by the 17-item Mental Health Inventory | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Menzies, PhD, APRN-BC, Principal Investigator — Florida International University
Locations (1):
- Florida International University, Miami, Florida, United States